CLINICAL TRIAL: NCT04602975
Title: A Phase 2a Age Descending Study to Investigate the Safety and Immunogenicity of the SF2a-TT15 Synthetic Carbohydrate-based Conjugate Vaccine Against Shigella Flexneri 2a in Adults, Children, and Infant Target Population in Endemic Countries.
Brief Title: A Study to Investigate the Safety and Immunogenicity of the SF2a-TT15 Synthetic Carbohydrate-based Conjugate Vaccine Against Shigella Flexneri 2a
Acronym: GlycoShig3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Wellcome Trust (Other); Gates Medical Research Institute (Other); Henry M. Jackson Foundation Medical Research International (Unknown); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); Parexel (Industry); ClinWin Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2018-017
Record Dates: First submitted 2020-09-24; First posted 2020-10-26 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: vaccine; anti-shigella; shigella; diarrheic disease; Kenya
MeSH Terms: conditions — Dysentery, Bacillary | interventions — Aluminum Hydroxide

STUDY DESIGN:
Intervention Model Description: Randomized, age descending (3 cohorts), with dose escalation in the target cohort
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Every team will be masked except the pharmacist and the pharmacy team on site and one dedicated personal within Sponsor team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Adults cohort 1 vaccinees (Experimental): Eligible subjects (adults - 18 to 50 yr-old) will be randomized to receive 3 intramuscular (IM) injections with the 10μg OS adjuvanted dose (or matching placebo), at a ratio of 3:1.
  Interventions: Biological: Injection SF2A-TT15 10 µg Adjuvanted
- Adults cohort 1 placebo recipients (Placebo Comparator): Eligible subjects (adults - 18 to 50 yr-old) will be randomized to receive 3 IM injections with the adjuvanted matching placebo.
  Interventions: Biological: Injection Adjuvanted Placebo
- Children cohort 2 vaccinees (Experimental): Eligible subjects (Children 2 to 5 yr-old) will be randomized to receive 3 IM injections of the 10 μg OS dose with Alhydrogel (or matching placebo) at a ratio of 3:1.
  Interventions: Biological: Injection SF2A-TT15 10 µg Adjuvanted
- Children cohort 2 placebo recipients (Placebo Comparator): Eligible subjects (Children 2 to 5 yr-old) will be randomized to receive 3 IM injections of the matching placebo with Alhydrogel.
  Interventions: Biological: Injection Adjuvanted Placebo
- Infants cohort 3A vaccinees (-) (Experimental): Eligible subjects (9 mo-old +/- 1mo infants) will be randomized to receive 3 IM injections of the not adjuvanted 2 μg dose (or of matching placebo), at a ratio of 4:1.
  Interventions: Biological: Injection SF2A-TT15 2 µg
- Infants cohort 3A placebo recipients (-) (Placebo Comparator): Eligible subjects (9 mo-old +/- 1mo infants) will be randomized to receive 3 IM injections of the not adjuvanted matching placebo.
  Interventions: Biological: Injection Placebo
- Infants cohort 3A vaccinees (+) (Experimental): Eligible subjects (9 mo-old +/- 1mo infants) will be randomized to receive 3 IM injections of the adjuvanted 2 μg dose (or of matching placebo), at a ratio of 4:1.
  Interventions: Biological: Injection SF2A-TT15 2 µg Adjuvanted
- Infants cohort 3A placebo recipients (+) (Placebo Comparator): Eligible subjects (9 mo-old +/- 1mo infants) will be randomized to receive 3 IM injections of the adjuvanted matching placebo.
  Interventions: Biological: Injection Adjuvanted Placebo
- Infants cohort 3B vaccinees (-) (Experimental): Eligible subjects (9 mo-old +/- 1mo infants) will be randomized to receive 3 IM injections of the not adjuvanted 10 μg dose (or of matching placebo), at a ratio of 4:1.
  Interventions: Biological: Injection SF2A-TT15 10 µg
- Infants cohort 3B placebo recipients (-) (Placebo Comparator): Eligible subjects (9 mo-old +/- 1mo infants) will be randomized to receive 3 IM injections of the not adjuvanted matching placebo.
  Interventions: Biological: Injection Placebo
- Infants cohort 3B vaccinees (+) (Experimental): Eligible subjects (9 mo-old +/- 1mo infants) will be randomized to receive 3 IM injections of the adjuvanted 10 μg dose (or of matching placebo), at a ratio of 4:1.
  Interventions: Biological: Injection SF2A-TT15 10 µg Adjuvanted
- Infants cohort 3B placebo recipients (+) (Placebo Comparator): Eligible subjects (9 mo-old +/- 1mo infants) will be randomized to receive 3 IM injections of the adjuvanted matching placebo.
  Interventions: Biological: Injection Adjuvanted Placebo

INTERVENTIONS:
Biological: Injection SF2A-TT15 10 µg Adjuvanted — Intramuscular injection of experimental vaccine (adjuvanted 10 µg)
  Other Names: SF2A-TT15 10 µg Adjuvanted; Anti-shigella experimental vaccine (10µg with alhydrogel)
  Arms: Adults cohort 1 vaccinees; Children cohort 2 vaccinees; Infants cohort 3B vaccinees (+)
Biological: Injection SF2A-TT15 10 µg — Intramuscular injection of experimental vaccine (not adjuvanted 10 µg)
  Other Names: SF2A-TT15 10 µg not adjuvanted; Anti-shigella experimental vaccine (10µg without alhydrogel)
  Arms: Infants cohort 3B vaccinees (-)
Biological: Injection Adjuvanted Placebo — Intramuscular injection of Placebo with alhydrogel
  Other Names: Placebo with Alhydrogel injection
  Arms: Adults cohort 1 placebo recipients; Children cohort 2 placebo recipients; Infants cohort 3A placebo recipients (+); Infants cohort 3B placebo recipients (+)
Biological: Injection Placebo — Intramuscular injection of the not adjuvanted Placebo
  Other Names: Placebo without alhydrogel injection
  Arms: Infants cohort 3A placebo recipients (-); Infants cohort 3B placebo recipients (-)
Biological: Injection SF2A-TT15 2 µg Adjuvanted — Intramuscular injection of experimental vaccine (adjuvanted 2 µg)
  Other Names: SF2A-TT15 2 µg Adjuvanted; Anti-shigella experimental vaccine (2µg with alhydrogel)
  Arms: Infants cohort 3A vaccinees (+)
Biological: Injection SF2A-TT15 2 µg — Intramuscular injection of experimental vaccine (not adjuvanted 2 µg)
  Other Names: SF2A-TT15 2 µg not adjuvanted; Anti-shigella experimental vaccine (2µg without alhydrogel)
  Arms: Infants cohort 3A vaccinees (-)

SUMMARY:
A study among adults, children and infants in Kenya to determine if a new type of glycoconjugate vaccine incorporating a synthetic carbohydrate component is safe and induces immunity against Shigella.

DETAILED DESCRIPTION:
The purpose of this study is to examine the safety and immunogenicity of two doses of the parenteral synthetic carbohydrate-based conjugate vaccine against Shigella flexneri 2a (Shigella flexneri 2a-Tetanus Toxoid15 (SF2a-TT15)) adjuvanted or not with Alhydrogel in infants in an endemic country (Kenya), the target population for the vaccine, using an age-descending approach. In total, 232 participants will be enrolled in the study: 16 adults (18-50 years-old), 16 children (2-5 years-old) and 200 infants (9 months-old +/ 1 mo).

The vaccine will be tested in adults first, then in children and eventually in infants in Kenya (where Shigella infection is present), based on the safety/tolerability in each group before to moving to the other. Participants will be randomly assigned to receive the study vaccine or a placebo control (same solution but without the vaccine component). The participants will have to go through all the trial procedures including the 14 visits (3 injections and 11 follow-up) during a 16 months period.

ELIGIBILITY:
Inclusion Criteria:

For adults:

1. Healthy men and women between 18 and 50 (inclusive) years of age.
2. Subjects who provide written informed consent or thumb print in the presence of a witness to participate in the study
3. Women willing to use at least 1 reliable method of contraception during the study period, or are surgically sterilized, and agree to undergo repeated pregnancy tests (before each vaccination) and men willing to use an effective method of contraception (e.g. condom).

For children and infants:

1. Healthy boys and girls between 2 and 5 years of age for the children group (cohort 2)
2. Healthy boys and girls 9 mo-old (+/- 1 month) for the infant group (cohort 3)
3. Parents or legally acceptable representatives, as appropriate, who are willing and able to provide signed/thumb printed informed consent for children and infants.
4. Infant and children should have a normal nutritional Z score (-2 or greater) according to the mother and child health handbook of the republic of Kenya - Ministry of Health before entering the trial.

For all:

1. Signed/thumb written informed consent, in accordance with local practice, provided by adult volunteers (participants 18 years of age and older), parent(s) or legal representative(s) for children and infants participants as applicable, who, in the opinion of the Investigator, can and will comply with the requirements of the protocol.
2. Subjects in general good health in the opinion of the Investigator as determined by medical history, vital signs and a physical examination.
3. No clinically significant abnormalities in hematology, blood chemistry, or urinalysis laboratory tests at screening.
4. Negative HIV, Hepatitis B and Hepatitis C serology tests and malaria test.

Exclusion Criteria:

1. Subjects with a history of clinically significant gastrointestinal disorders (e.g. gastroesophageal reflux disease, peptic ulcer, celiac disease, inflammatory bowel disease).
2. Individuals with immunosuppressive diseases or under immunosuppressive therapy.
3. Previous participation in any study in which a Shigella-vaccine candidate was administered.
4. Suspected or known hypersensitivity (including allergy) to any of the vaccine components or to previous vaccine, or to medicinal products or medical equipment whose use is foreseen in this study.
5. Use of any prescription or over-the-counter (OTC) medications, within 14 days prior vaccination. Paracetamol or ibuprofen for symptomatic relief of pain is allowed until 48 hours prior to vaccination.
6. Women who are pregnant, breast-feeding, or are of childbearing age and are not on or do not plan to use acceptable contraceptives for the duration of the study.
7. Subjects with any significant acute medical situation (e.g. acute infection) within 48 hrs prior to study entry, in the opinion of the Principal Investigator.
8. Participation in another clinical trial with drugs within 3 months prior first study injection.

Ages: 8 Months to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 248 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Number, proportion,severity and relatedness of adverse events (AEs) to measure the safety and tolerability of SF2a-TT15 vaccine (2 μg OS and 10 μg OS) in each cohort. | 15 months
  Solicited reactions, AEs, SAEs assessed post-vaccination using targeted physical examinations, vital signs, and clinical laboratory tests
Analyses of the serum anti-S. flexneri 2a lipopolysaccharide (LPS) IgG antibody response in the infant target population to assess the immunogenicity of the vaccine. | 15 months
  Proportion of responders (4-fold increases over baseline) in serum anti-S. flexneri 2a LPS IgG antibody response

SECONDARY OUTCOMES:
The number and proportion of responders, the geometric mean titer (GMT), mean fold-rises (compared to baseline), and peak-post-vaccination of the serum bactericidal activity (SBA) antibody (functionality of SF2a-specific IgGs antibodies in infants). | 15 months
  Proportion of responders (4-fold increases over baseline) in serum bactericidal activity (SBA) antibody
Analyses of the serum anti-S. flexneri 2a LPS Immunoglobulins G (IgG) antibody response in the adult and children cohorts. | 15 months
  Proportion of responders (4-fold increases over baseline) in serum anti-S. flexneri 2a LPS IgG antibody response
Comparison of the Measle-Rubella (MR) vaccine immune response in SF2a-TT15 vaccinees and placebo groups for the infant cohort. | 15 months
  The antibody titer to the MR vaccine will be compared between SF2a-TT15 vaccinees and placebo groups to assess whether the SF2a-TT15 Shigella vaccine candidate impacts on the immunogenicity of the MR vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Armelle Phalipon, PhD, Study Chair — Institut Pasteur; Laurence Mulard, PhD, Study Chair — Institut Pasteur; Christiane Gerke, PhD, Study Chair — Institut Pasteur (Consulting); Fredrick Sawe, MBChB MMED, Principal Investigator — Kenya Medical Research Institute
Locations (1):
- KEMRI / Henry M. Jackson Foundation Medical Research International, Kericho, Kenya

IPD SHARING:
Plan to Share IPD: No
This study is a part of a development program, Data will stay confidential and possibly shared only with program partners.